CLINICAL TRIAL: NCT03382717
Title: Clinical Evaluation of Efficacy and Safety of a Medical Device for the Treatment of Toenail Onychomycosis.
Brief Title: Efficacy and Safety of a Medical Device for the Treatment of Toenail Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16E1078
Record Dates: First submitted 2017-12-11; First posted 2017-12-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Onychomycosis of Toenail

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Excilor Forte (Experimental): One application of the MD daily (at same time point), preferably after showering/bathing, during the complete study period.
  Interventions: Device: Excilor Forte
- Loceryl 5% (Active Comparator): One application per week of the positive control Loceryl 5% during the whole study period.
  Interventions: Drug: Loceryl 5%

INTERVENTIONS:
Device: Excilor Forte — 1 application per day during 6 months
  Arms: Excilor Forte
Drug: Loceryl 5% — 1 application per week during 6 months
  Arms: Loceryl 5%

SUMMARY:
This study evaluates the effect of the medical device "Excilor® Forte" in the treatment of toenail onychomycosis. Half of the participants will receive the tested product and the other half will receive a comparator (Amorolfin 5%). Patients will be followed during 6 months.

DETAILED DESCRIPTION:
Subjects with a great toenail, affected by onychomycosis, were treated with the test medical device or reference product, respectively. After 180 days, blind assessment of the % of healthy surface (primary end point) of the great toenail was performed to compare the effect of both treatments, and to evaluate improvement versus baseline (day 0), respectively. Additionally, blind assessment of the percentage of healthy surface of the great toenail was performed at all other visits (D30, D60, D120) to evaluate changes from baseline between both treatment groups. For this purpose, digital macrophotographs were analysed by a blinded investigator using Adobe Photoshop software.

ELIGIBILITY:
Inclusion Criteria:

* Subject having given her/his informed, written consent.

  * Subject cooperative and aware of the modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.
  * Subject being psychologically able to understand information and to give their/his/her consent.
  * Age: more than 18 years.
  * Subject with superficial onychomycosis on at least one great toenail or light to moderate disto-lateral onychomycosis (without matrix involvement and involvement <2/3 of the tablet).
  * Subject with positive KOH staining.
  * Subject having stopped any systemic antifungal treatment since at least 6 months before inclusion and/or any topical antifungal treatment since at least 3 months before inclusion.
  * Female subjects of childbearing potential should use an accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after study end.

Exclusion Criteria:

* Subject considered by the Investigator likely to be non-compliant with the protocol.
* Patient enrolled in another clinical trial during the test period.

  · Woman being pregnant, nursing or planning a pregnancy during the course of this study.
* Subject having a known allergy to one of the constituents of the tested products.
* Patient suffering from serious or progressive diseases (to investigator's discretion) such as uncontrolled diabetes, peripheral circulatory disease, HIV, psoriasis, lichen planus, immunosuppressive pathology…
* Subject with cutaneous pathology on studied zone (other than onychomycosis like angioma, dermatitis…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2017-08-26 (Actual); Study Completion 2017-08-26 (Actual)

PRIMARY OUTCOMES:
Variation of the percentage of healthy surface after 30, 60, 120, and 180 days between both treatments, and versus baseline. Evaluation is done by digital analysis of photographs of the great, infected toenail | After 30, 60, 120 and 180 days of treatment
  Subjects with a great toenail, affected by onychomycosis, were treated with the test medical device or reference product, respectively. After 180 days, blind assessment of the percentage of healthy surface (primary efficacy endpoint) of the great toenail was performed to evaluate changes from baseline between both treatment groups. Additionally, blind assessment of the percentage of healthy surface of the great toenail will be performed at all other visits (day 30, 60, and 120, respectively) to evaluate changes from baseline between both treatment groups

SECONDARY OUTCOMES:
Evaluation of clinical efficacy by the investigator, assessing the following parameters: onychomycosis evolution, onycholysis, dystrophy, discoloration, and nail thickening, following treatment with test medical device versus reference product. | After 30, 60, 120 and 180 days of treatment
  Onycholysis, nail distrophy, nail discoloration, and nail thickening was evaluated by a blinded investigator, using the following scores: 0 = none, 1 = very slight, 2 = slight, 3 = moderate, and 4 = severe. Onychomycosis evolution was scored as follows: 1 = failure (aggravation, increase total infected area), 2 = status quo, 3 = improvement (decrease of total infected area), 4 = success: disappearance of the total infected area. In order to compare changes in nail dystrophy, discoloration, and nail thickening between baseline and day 180, five categories were reduced to two categories (none to slight versus moderate to severe). The Mc Nemar test for paired data was used to test if there was a change in nail dystrophy, discoloration, and nail thickening between baseline and day 180. A chi-square test test was performed to compare changes between both treatments in onychomycosis evolution.
  Note: scores are used and for this reason, no units of measure can be assigned.
Evaluation of microbiological efficacy of the product, using KOH staining and fungal culture on D0 and D180 versus reference product. | At baseline (day 0) and after 180 days of treatment
  Patients with positive KOH staining were included in the study. In addition, a fungal culture was performed to identify the involved species. At day 180, a new KOH staining and fungal culture was performed to evaluate the impact of each treatment on both microbiological parameters.
Evaluation of product tolerance at each visit during the trial, assessed by the investigator by clinical evaluation and subject interrogatory. | After 30, 60, 120 and 180 days of treatment
  The investigator assigned a score from 0 (bad tolerance) to 3 (very good tolerance).
Evaluation of the quality of life of the subjects using a validated questionnaire (NailQoL) before (baseline), after 60 and 180 days of treatment with test product, versus comparator. | After 60 and 180 days of treatment
  A NailQol global score of 0 corresponds with a quality of life never altered by onychomycosis, whereas a score of 100 corresponds to a quality of life that is always affected by onychomycosis.
Subject evaluation using an evaluation questionnaire, performed at each visit. | After 30, 60, 120 and 180 days of treatment
  A questionnaire was included to evaluate product usability and functionality of Excilor Forte. The questionnaire was completed at each evaluation point (day 30, 60, 120, and 180, respectively). General questions were asked regarding the cosmetic effect (e.g. smoothening, brightening effect, conventional packaging..), overall satisfaction (e.g. smell, fits daily routine ...), product application (e.g. ease of application, drying time, stress-resistance, combination with top coat...), purchase intent and tolerance were asked. Subjects needed to score as follows: strongly agree, agree, neutral, disagree, strongly disagree, not concerned. Data were summarized in frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Nejib Doss, MD, Principal Investigator — Principal Instruction military hospital of Tunis
Locations (2):
- Tunisia (2):
  - Hospital Habib Thameur, Tunis
  - Principal instruction military hospital, Tunis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eertmans F, Doss N, Rossel B, Adriaens E. Daily Application of an Aqueous, Acidifying, Peelable Nail Polish versus Weekly Amorolfine for Topical Onychomycosis Treatment: A Prospective, Randomized, Blinded Trial. Dermatol Ther (Heidelb). 2018 Sep;8(3):463-473. doi: 10.1007/s13555-018-0254-1. Epub 2018 Jul 26. PMID 30051298